CLINICAL TRIAL: NCT02453815
Title: Do Arterial Catheters Reduce the Risk of Major Perioperative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-008
Record Dates: First submitted 2015-02-12; First posted 2015-05-27 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- arterial catheter (Experimental): If a patient is randomized by the web-based system before non-cardiac surgery to receive an arterial catheter at surgery, then the subject will be placed in the experimental arm of the study.
  Interventions: Procedure: non-cardiac surgery; Other: arterial catheter
- no arterial catheter (Placebo Comparator): If a patient is randomized by the web-based system before non-cardiac surgery to not receive an arterial catheter at the time of surgery, then the subject will be placed in the placebo comparator arm of the study.
  Interventions: Procedure: non-cardiac surgery

INTERVENTIONS:
Procedure: non-cardiac surgery — all surgical procedures except cardiac
Other: arterial catheter — arterial catheter
  Arms: arterial catheter

SUMMARY:
Even slight reduction in serious complications related to blood pressure management would easily justify the cost and relatively rare complications consequent to arterial catheter insertion. However, it seems unlikely that major outcomes will be improved by the presumably slight difference in hemodynamic control resulting continuous blood pressure measurement rather than measurements at 2-5-minute intervals. There is considerable variation in practice and no clear consensus whether arterial lines should be placed or not, especially in ASA 2 patients undergoing major non-cardiac surgery or ASA-3 patients undergoing moderate to major non-cardiac surgery. Clearly, if there is no benefit to outcome, arterial lines, which are invasive and costly, should not be placed routinely. The investigators therefore propose to test the primary hypothesis that use of arterial catheters decreases the risk of a collapsed composite of in-hospital mortality, re-admissions, MINS, AKI, stroke, respiratory and wound healing and gastro-intestinal complications after non-cardiac surgery.

Secondarily, the investigators propose to test the hypotheses that arterial catheter use: 1) decreases the duration of hospitalization; 2) increases blood gas, electrolyte, and coagulation testing; 3) increases induction-to-incision time; and, 4) increases cost-of-care (supplies,, blood tests, and induction-to-incision time).

DETAILED DESCRIPTION:
This study will be conducted at the Cleveland Clinic Main Campus with IRB approval and written consent from participating patients. The investigators will enroll consented ASA Physical Status 2-4 patients having inpatient non-cardiac surgery in whom a radial arterial catheter might or might not reasonably be used based on co-morbidity or type of surgery. However, it is most likely that the majority of patients will be ASA 3 patients. Currently (based on a recent data pull) approximately 44% of ASA 3 patients receive an arterial catheter for non-cardiac surgery. The investigators expect that this insertion rate will remain constant throughout the study.

Aside from randomized assignment to arterial catheter use, no other aspect of anesthetic or perioperative management will be controlled.

When attending anesthesiologists exclude otherwise qualifying patients from the study, the investigators will ask them to designate which factors influenced their decision. Potential reasons will include: 1) type of procedure; 2) co-morbidities; 3) expected hemodynamic instability or blood loss; 4) patient position; and, 5) need for blood sampling.

Demographic data to be obtained includes height (cm), weight (kg), age (yr.), gender, ASA physical status, and self-declared ethnicity. If available the investigators will collect social history (tobacco and alcohol use), medical history (pulmonary disease, cardiovascular disease, neurologic disease, drug usage (including but not limited to: statins, ß blockers, oral hypoglycemic agents and/or insulin), NSAIDs, diabetes (and whether insulin-dependent or not), and previous glucose-tolerance test results, preoperative hemoglobin and hematocrit, BUN and creatinine, electrolytes, preoperative EKG, and hemoglobin A1c (HbA1c).

Anesthetic data will include volatile anesthetic dose in MAC-hours, as well as total doses of propofol and other sedative hypnotics. Hemodynamic, respiratory parameters, BIS values (if available) and distal esophageal temperature will be recorded at 10 minute intervals intraoperatively. Blood loss will be estimated; urine output and fluid administration including allergenic blood will be recorded. Intraoperative use and total dose of vasoactive drugs as well as antibiotic administration will be recorded. The investigators will also record duration of anesthesia as well as time from induction of anesthesia to surgical incision. Similar data will be recorded for patients who potentially qualify but are excluded from randomization by the attending anesthesiologist.

Serum troponin and creatinine will be determined on postoperative days 1, 2 and 3 while in hospital. Blood will be drawn in conjunction with routine laboratory tests. The surgical team will be notified when troponin values ≥0.03 ng/ml are identified.

All other study data will be obtained from the medical record, including patient characteristics, type of surgery, perioperative blood transfusions, mean-arterial pressure, vasopressor use, number of blood gas and coagulation tests, and duration of hospitalization, postoperative complications as well as readmissions.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 2-4 patients
* inpatient non-cardiac surgery
* radial arterial catheter might or might not reasonably be used based on co-morbidity or type of surgery.

Exclusion Criteria:

* the attending anesthesiologist requires or refuses an arterial catheter
* already have an arterial catheter
* catheter is contraindicated
* end-stage renal disease
* abnormal Allen's test
* known radial arterial pathology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2015-06; Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Number of post operative complications | 30 days
  Medical record will be reviewed for number of post operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States